CLINICAL TRIAL: NCT01123564
Title: A Randomized, Controlled, Two-center Phase II Study Assessing the Efficacy and Safety of Intravitreal Lucentis Injections in Patients With Clinically Significant Macular Edema Secondary to Central Retinal Vein Occlusion
Brief Title: Efficacy and Safety of Lucentis for Clinically Significant Macular Edema Secondary to Central Retinal Vein Occlusion
Acronym: BRAVO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pecs (Other)
Collaborators: University of Debrecen (Other)
Responsible Party: Zsolt Balla/assistant lecturer, University of Pecs, Medical Scool, Dept of Ophthalmology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002AHU02T
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Retinal Vein Occlusion; Macular Edema
Keywords: macular edema secondary to retinal vein occlusion
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lucentis (ranibizumab) (Experimental)
  Interventions: Drug: ranibizumab
- Laser (Active Comparator)
  Interventions: Radiation: Argon laser treatment

INTERVENTIONS:
Drug: ranibizumab — applied monthly in the first 3 months period, and after this only if visual acuity (VA) decreases with more than 5 letters at any monthly visits
  Other Names: Lucentis intravitreal injection
  Arms: Lucentis (ranibizumab)
Radiation: Argon laser treatment — Conventional grid pattern argon laser treatment and panretinal argon laser photocoagulation in an as needed basis.
  Other Names: Laser photocoagulation
  Arms: Laser

SUMMARY:
This study aims to assess if Lucentis injection applied into the eye is superior to conventional treatment concerning the prevention of visual loss in patients having clinically significant macular edema secondary to retinal vein occlusion

ELIGIBILITY:
Inclusion Criteria:

* Macular edema persisting for more than 3 months period despite conventional medication.
* Central retinal vein occlusion is confirmed by slit-lamp biomicroscopy and fluorescein angiography (FLAG).
* Patients randomized into ranibizumab-treated group do not receive macular laser treatment.
* Macular edema is defined by OCT: the thickness of central foveal area calculated by macular map analysis is above 280 μm and/or retinal thickness is above 330 μm at any region of the macula calculated by retinal thickness analysis.
* Baseline visual acuity is less than 64 ETDRS letters (or 0.4 decimal equivalent).

Exclusion Criteria:

* Diabetes mellitus
* Additional vitreoretinal diseases
* History of pars plana vitrectomy
* Previous macular grid laser treatment
* Intravitreal triamcinolone acetonid treatment
* Complicated cataract surgery
* Advanced glaucomatous damage of optic nerve head
* Cataract (except mild, defined as grade 1 nuclear sclerosis and/or grade 1 posterior subcapsular cataract)
* Age-related macular degeneration
* Pregnancy and lactation
* Women in childbearing potential who are not using double safe contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy compared to conventional treatment assessed by BCVA(best corrected visual acuity) | 12 months
  To assess the superiority of intravitreal (IVT) ranibizumab to conventional treatment concerning prevention of visual loss or improvement of BCVA as determined by the mean change of BCVA tested by ETDRS chart compared to baseline in 12 months period, when intravitreal ranibizumab is applied monthly in the first 3 months period, and later when visual acuity (VA) decreases with more than 5 letters at any visit performed monthly.

SECONDARY OUTCOMES:
Efficacy assessed by change in macular thickness | 12 months with monthly assessment
  The efficacy of treatment concerning change of anatomical structure of macular region detected by Optical Coherence Tomography (OCT) - the mean change of macular thickness (micron) at each months of 1 year period.

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Balla, MD PhD, Principal Investigator — University of Pecs
Locations (2):
- Hungary (2):
  - Debrecen Medical and Health Science Center Dept of Ophthalmology, Debrecen
  - University of Pecs, Medical School, Department of Ophthalmology, Pécs